CLINICAL TRIAL: NCT04252625
Title: A Phase II Randomized Controlled Trial of a Supplement Containing Quercetin, Bromelain, Rye Flower Pollen, and Papain on Reducing the Severity of Radiation-Induced Prostatitis
Brief Title: Trial of Quercetin, Bromelain, Rye Flower Pollen & Papain on Reducing Severity of Radiation-Induced Prostatitis
Acronym: Q-Urol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug Supply Issue
Sponsor: University of Utah (Other)
Collaborators: Farr Labs, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCI129154
Record Dates: First submitted 2020-01-23; First posted 2020-02-05 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: An asymmetric two-sided group sequential design will be used with an interim analysis for efficacy and futility.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Q-Urol (Active Comparator): Patients will be randomized in a 1:1 ratio to receive Q-Urol, two capsules, twice daily for 6 weeks after brachytherapy placement.
  Questionnaires will be administered pre- and post-treatment to assess the change in prostatitis symptoms and quality of life measures. The mean values between groups will be compared.
  Interventions: Drug: Q-Urol
- Arm 2: Placebo (Placebo Comparator): Patients will be randomized in a 1:1 ratio to receive Placebo, two capsules, twice daily for 6 weeks after brachytherapy placement.
  Questionnaires will be administered pre- and post-treatment to assess the change in prostatitis symptoms and quality of life measures. The mean values between groups will be compared.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Q-Urol — Q-Urol is an over-the-counter herbal supplement manufactured by Farr Laboratories. It is a combination product composed of quercetin, pollen extract, bromelain, and papain.
  Arms: Arm 1: Q-Urol
Drug: Placebo — placebo capsule
  Arms: Arm 2: Placebo

SUMMARY:
This study will assess the difference in prostatitis symptoms in men with localized prostate cancer following brachytherapy taking Q-Urol relative to placebo.

DETAILED DESCRIPTION:
This is a Phase 2, double-blinded, placebo-controlled trial assessing the safety of Q-Urol use after brachytherapy placement in patients with localized prostate cancer. Patients will be randomized in a 1:1 ratio to receive Q-Urol/Placebo twice daily for 6 weeks after brachytherapy placement. Questionnaires will be administered pre- and post-treatment to assess the change in prostatitis symptoms and quality of life measures. The mean values between groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged ≥ 18 years.
* Men with histologically proven localized prostate adenocarcinoma, stage I - III (as defined by American Joint Committee on Cancer (AJCC) 8th edition), who have selected treatment with brachytherapy with or without external beam radiation, with or without androgen deprivation therapy.
* Fluent in speaking and reading English.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
* Adequate organ function as defined as:

  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
    * aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 × institutional ULN
  * Renal:

    * Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula:

      * Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
* Highly effective contraception for both male and their female partners of childbearing potential throughout the study and for at least 5 days after last study treatment administration if the risk of conception exists.
* Median life expectancy ≥ 5 years as calculated by the Lee and Schonberg Index (https://eprognosis.ucsf.edu/leeschonberg.php)
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Baseline AUA symptom scores > 15.
* Prior diagnosis of chronic prostatitis type II through IV.
* Subject has received systemic therapy intended for the treatment of prostatitis (including herbal supplements) ≤ 14 days of starting study treatment.
* Subject has received a fluoroquinolone antibiotic (e.g. ciprofloxacin, norfloxacin, ofloxacin levofloxacin, etc.) ≤ 3 days of starting study treatment.
* Subject is actively on anti-inflammatory medications for other medical conditions, unless approved by PI.
* Subject has undergone transurethral resection of the prostate (TURP).
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* History of irritable bowel syndrome, chronic fatigue syndrome, fibromyalgia, and interstitial cystitis-bladder pain syndrome (IC/BPS).
* History of symptomatic hypotension, falls, or syncope
* History of hypoglycemia.
* Actively abusing alcohol or drugs
* Subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Congestive heart failure
  * Diabetes
  * Pulmonary artery hypertension
  * Any clinically significant condition that requires therapy with diuretic medications for any indication other than the management of hypertension.
  * Other clinically significant disorders that would, in the opinion of the treating investigator, preclude safe study participation.
* Known prior severe hypersensitivity to investigational product or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Known allergy to pineapple or pineapple containing products.
* Subjects taking prohibited medications as described in Section 7.3 A washout period of prohibited medications for a period of at least 5 half-lives or as clinically indicated should occur prior to the start of treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male subjects ≥ 18 years
Enrollment: 10 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tward, MD, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (2):
- United States (2):
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Q-Urol: Patients were randomized in a 1:1 ratio to receive Q-Urol, two capsules, twice daily for 6 weeks after brachytherapy placement.
  Questionnaires were administered pre- and post-treatment to assess the change in prostatitis symptoms and quality of life measures. The mean values between groups will be compared.
  Q-Urol: Q-Urol is an over-the-counter herbal supplement manufactured by Farr Laboratories. It is a combination product composed of quercetin, pollen extract, bromelain, and papain.
- Arm 2: Placebo: Patients were randomized in a 1:1 ratio to receive Placebo, two capsules, twice daily for 6 weeks after brachytherapy placement.
  Questionnaires were administered pre- and post-treatment to assess the change in prostatitis symptoms and quality of life measures. The mean values between groups will be compared.
  Placebo: placebo capsule
Period: Overall Study
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.60 (6.88) | 64.00 (7.81) | 63.30 (6.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI)
Description: This outcome will report the mean score of the NIH-CPSI, a 13-item questionnaire.
  This questionnaire will report 4 sub-scores, Pain, Urinary Symptoms, Quality of Life (QOL) Impact, and Pain + Urinary score, and the total score.
  Pain: The sum of 6 items (0 No-1 Yes), one scale (0 Never-5 Always), and one scale (0 No Pain-10 Pain as bad as you can imagine); Range: 0-21, higher values indicating worse outcomes.
  Urinary Symptoms: The sum of 2 urine items (0 Not at all-5 Almost always); Range: 0-10, higher values indicating worse outcomes.
  QOL Impact: The sum of 2 items (0 None-3 A lot) and 1 scale (0 Delighted-6 Terrible); Range: 0-12, higher values indicating worse outcomes.
  Pain and Urinary sub-score: The sum of the Pan and Urinary Symptoms scores; Range: 0-31, higher values indicating worse outcomes.
  Total Score: The sum of all questions; Range: 0-43, higher values indicating worse outcomes.
  This outcome measure is assessed at 6 weeks after the start of study treatment.
Time Frame: up to 6 weeks after the start of study treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm 1: Q-Urol: Patients were randomized in a 1:1 ratio to receive Q-Urol, two capsules, twice daily for 6 weeks after brachytherapy placement.
  Questionnaires were administered pre- and post-treatment to assess the change in prostatitis symptoms and quality of life measures. The mean values between groups were compared.
  Q-Urol: Q-Urol is an over-the-counter herbal supplement manufactured by Farr Laboratories. It is a combination product composed of quercetin, pollen extract, bromelain, and papain.
- Arm 2: Placebo: Patients were randomized in a 1:1 ratio to receive Placebo, two capsules, twice daily for 6 weeks after brachytherapy placement.
  Questionnaires were administered pre- and post-treatment to assess the change in prostatitis symptoms and quality of life measures. The mean values between groups were compared.
  Placebo: placebo capsule
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Number analyzed (Participants) | 5 | 5
score on a scale
  Pain Score | 4.00 (4.24) | 5.8 (4.27)
  Urinary Symptoms Score | 6.00 (2.55) | 4.60 (2.51)
  Quality of life impact Score | 4.80 (1.30) | 5.20 (2.59)
  Pain score and urinary Score | 10 (5.24) | 10.4 (5.13)
  Total Score | 14.80 (6.38) | 15.60 (7.09)

2. Secondary Outcome: The Expanded Prostate Cancer Index Composite (EPIC) Assessment
Description: Health Related Quality of Life (HRQOL) will be assessed with EPIC questionnaires. Items are standardized to a 0-100 scale and are averaged to calculate four subscale scores (Urinary Summary, Bowel Summary, Sexual Summary, Hormonal Summary). A higher score (max 100) represents better HRQOL, and a lower score (min 0) represents worse HRQOL.
Time Frame: up to 6 weeks after the start of study treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Number analyzed (Participants) | 5 | 4
score on a scale
  Urinary Summary | 68.62 (10.89) | 64.44 (15.87)
  Bowel Summary | 85.36 (12.01) | 84.37 (11.42)
  Sexual Summary | 26.44 (40.81) | 23.71 (17.22)
  Hormonal Summary | 72.02 (17.81) | 75.03 (12.42)

3. Secondary Outcome: The International Prostate Symptom Score (I-PSS) Assessment
Description: Health Related Quality of Life (HRQOL) will be assessed with International Prostate Symptom Score (I-PSS). This is a questionnaire with 7 questions concerning urinary symptoms (from 0 to 5). A high score (max 35) indicates worse HRQOL and a low score (min 0) represents a better HRQOL. These score are reported as Mild (0-7), moderate (8-19) or Severe (20-35).
  total score ranges from 0 to 35 (asymptomatic to very symptomatic).
Time Frame: up to 6 weeks after the start of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Number analyzed (Participants) | 5 | 5
Participants
  Mild | 0 | 0
  Moderate | 2 | 4
  Severe | 3 | 1

4. Secondary Outcome: The Rectal Function Assessment Score (R-FAS) Assessment
Description: Health Related Quality of Life (HRQOL) will be assessed with the R-FAS 10-item questionnaires. Question 10 does not count toward the total score. 9 questions are scored from 0-3. A higher score represents poorer bowel function (max 27) and a lower score represents better bowel function (min 0).
Time Frame: At the End of Treatment Visit, up to 8 weeks after initiation of study treatment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Number analyzed (Participants) | 5 | 5
Score on a scale | 5.20 (2.95) | 3.60 (3.36)

5. Secondary Outcome: Sexual Health Inventory for Men (SHIM) Assessment
Description: The SHIM is a 5 point questionnaire with ratings from 0-5 to assess Health Related Quality of Life (HRQOL). The sum of the SHIM score is categorized to Severe Erectile Dysfunction ED (0-7), Moderate ED (8-11), Mild to Moderate ED (12-16), Mild ED (17-21), No signs of ED (22-25).
  This outcome will report the count of participants in each category.
Time Frame: At the End of Treatment Visit, up to 8 weeks after initiation of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Number analyzed (Participants) | 5 | 5
Participants
  Severe Erectile Dysfunction ED (0-7) | 3 | 3
  Moderate ED (8-11) | 0 | 1
  Mild to Moderate ED (12-16) | 0 | 0
  Mild ED (17-21) | 0 | 1
  No signs of ED (22-25) | 1 | 0
  Not assessed | 1 | 0

6. Secondary Outcome: Impact on Serum Biomarkers of Inflammation - Erythrocyte Sedimentation Rate (ESR)
Description: The inflammation marker, erythrocyte sedimentation rate (ESR), was collected at the End of Treatment visit for comparison between treatment and placebo groups. This outcome will report the mean ESR of each arm.
Time Frame: At the End of Treatment Visit, up to 8 weeks after initiation of study treatment.
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Number analyzed (Participants) | 4 | 4
mm/hour | 4.50 (1.73) | 2.50 (1.73)

7. Secondary Outcome: Impact on Serum Biomarkers of Inflammation - C-reactive Protein
Description: The inflammation marker, C-reactive protein, was collected at the End of Treatment visit for comparison between treatment and placebo groups.
  This outcome will report the mean C-reactive protein of each arm.
Time Frame: At the End of Treatment Visit, up to 8 weeks after initiation of study treatment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Number analyzed (Participants) | 5 | 4
mg/dL | 0.14 (0.11) | 0.48 (0.62)

8. Secondary Outcome: Impact on Serum Biomarkers of Inflammation - Prostate-specific Antigen (PSA)
Description: The inflammation marker, Prostate-specific antigen (PSA), was collected at the End of Treatment visit for comparison between treatment and placebo arm.
  This outcome will report the mean PSA of each arm.
Time Frame: At the End of Treatment Visit, up to 8 weeks after initiation of study treatment.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Number analyzed (Participants) | 5 | 4
ng/ml | 1.11 (0.90) | 1.87 (0.92)

9. Secondary Outcome: Adverse Events by Grade
Description: To assess safety of Q-Urol compared to placebo. The severity of adverse events was assessed using CTCAE v5.0 criteria, a 1-5 scale with higher numbers indicating greater severity. Grade 1 indicates "mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated" and Grade 5 indicates "death related to AE".
  This outcome measure will report the following:
  The count of participants who had a grade 1-2 event, related to study treatment.
  The count of the participants who had a grade 3-4 event, related to study treatment.
  The count of the participants who had a grade 5 event or higher.
  Subjects were monitored for adverse events from the start of treatment until 30 days after the last dose of study treatment.
Time Frame: up to 10.5 weeks after initiation of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Number analyzed (Participants) | 5 | 5
Participants
  Grade 1-2 | 5 | 5
  Grade 3-4 | 0 | 0
  Grade 5 | 0 | 0

10. Secondary Outcome: Days of Pain Medication
Description: To assess effect on prostatitis-related pain in men with localized prostate cancer following brachytherapy taking Q-Urol relative to placebo. This outcome will report the mean number of days participants took pain medication as documented on a self reported Pain Management Diary. This was followed for 28 days; the minimum number of days is 0 and the maximum number is 28.
Time Frame: up to 28 days after initiation of study treatment
Measure: Mean (Standard Deviation); unit: Pain Medication days
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
Number analyzed (Participants) | 5 | 5
Pain Medication days | 6.00 (6.75) | 5.20 (6.30)

ADVERSE EVENTS:
Time Frame: The collection of adverse events, serious adverse event, and survival began after the study drug was started and ended 30 days after the last dose study drug (or until new cancer treatment was initiated), up to 13 weeks after treatment initiation.
Arm/Group | Arm 1: Q-Urol | Arm 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Q-Urol (N=5) | Arm 2: Placebo (N=5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 2 (3)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (4) | 2 (2)
Pain (General disorders) | 2 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 1 (2)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Weight loss (Investigations) | 1 (2) | 2 (3)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04252625/Prot_SAP_000.pdf